CLINICAL TRIAL: NCT06862284
Title: Efficacy, Safety and Immunological Effect of Upadacitinib in the Treatment of Primary Sjögren's Syndrome
Brief Title: Therapeutic Effect of Upadacitinib in Primary Sjögren's Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, He Jing, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pss2024upa
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-12

CONDITIONS: Primary Sjögren's Syndrome (pSS)
MeSH Terms: interventions — upadacitinib; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- upadacitinib group (Experimental): Participants will receive upadacitinib 15 milligrams (mg) orally once daily for 52 weeks.
  Interventions: Drug: Upadacitinib (ABT-494)
- hydroxychloroquinone group (Active Comparator): Participants will receive hydroxychloroquine 200 milligrams (mg) orally twice daily for 52 weeks.
  Interventions: Drug: Hydroxychloroquine (HCQ)

INTERVENTIONS:
Drug: Upadacitinib (ABT-494) — Upadacitinib 15mg Qd for 52 weeks
  Arms: upadacitinib group
Drug: Hydroxychloroquine (HCQ) — Hydroxychloroquine 200mg Bid for 52 weeks
  Arms: hydroxychloroquinone group

SUMMARY:
This study is designed to explore the efficacy and safety of upadacitinib and clarify the influence on immune function in the treatment of primary Sjögren's Syndrome.

DETAILED DESCRIPTION:
This is an open-label, single-center, randomized controlled trial of upadacitinib in the treatment of active primary Sjögren's Syndrome. The enrollment was based on the American College of Rheumatology(ACR) and European League Against Rheumatism (EULAR)(2016) diagnostic criteria. The efficacy and safety were evaluated in participants given upadacitinib 15mg/day and a proper, stable dose of hydroxychloroquine 400mg/day. Changes in clinical manifestation, laboratory indexes, and immunological indicators were explored in the process.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >18 years of age at screening visits
2. Participants with diagnosis of pSS according to the 2016 ACR/EULAR criteria
3. Participants have an ESSDAI score ≥ 5
4. Participants must be on a stable dose of prednisone (≤10mg/day), antimalarials or equivalent, and cholinergic stimulants prior to Baseline.
5. Participants previously on other immunosuppressive drugs (methotrexate, azathioprine, mycophenolate mofetil, cyclosporine, tacrolimus, iguratimod) should have withdrawn drug for at least 8 weeks (56 days) at the time of screening
6. If the subject has evidence of new latent tuberculosis (TB) infection, the subject must initiate and complete a minimum of 2 weeks (or per local guidelines, whichever is longer) of an ongoing TB prophylaxis before continuing to receive the study drug.
7. If female, the subject must be postmenopausal, OR permanently surgically sterile, OR for women of childbearing potential practicing at least one protocol-specified method of birth control, that is effective from Study Day 1 through at least 30 days after the last dose of study drug.
8. The patient must be informed in writing of the consent to participate in the trial and the patient is expected to be able to comply with the requirements of the study follow-up plan and other protocols.

Exclusion Criteria:

Any subject meeting any of the following criteria should be excluded:

1. Pregnant or breastfeeding female.
2. Diagnosis of other autoimmune disease, or other sicca syndrome.
3. Laboratory value abnormality:

(1)Serum aspartate transaminase (AST) or alanine transaminase (ALT) > 3.0 × upper limit of normal (ULN); (2)Estimated glomerular filtration rate by simplified 4-variable Modification of Diet in Renal Disease (MDRD) formula < 40 mL/min/1.73m^2; (3)Total white blood cell count (WBC) < 2,000/μL; (4)Absolute neutrophil count (ANC) < 1,000/μL; (5)Platelet count < 50,000/μL; (6)Absolute lymphocytes count < 500/μL; (7)Hemoglobin < 8 g/dL.

4. Ongoing infections at Week 0 that have not been successfully treated.

5. Infection with HIV ( HIV antibody positive serological test ) or hepatitis C ( hepatitis C antibody positive serological test ). If the serum reaction is positive, it is recommended to consult a doctor with expertise in the treatment of HIV or hepatitis C virus infection.

6. History of any known malignancy in the last 5 years (except non-melanoma skin cancer, non-melanoma skin cancer or cervical tumors that have not recurred within 3 months after surgical cure prior to screening).

7. Underlying cardiac, pulmonary, metabolic, renal, hepatic, gastrointestinal, hematological or neurological conditions, chronic or latent infectious diseases, or immune deficiency which places the patient at an unacceptable risk for participation in the study.

8. Prior exposure to any Janus kinase (JAK) inhibitor (including but not limited to tocilizumab, sirukumab, sarilumab, upadacitinib, tofacitinib, baricitinib, ruxolitinib, peficitinib, and filgotinib).

9. Exposure to biological DMARDs in two months before screening.

10. Enrollment in another interventional clinical study while participating in this study.

11. Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive the study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Treatent response assessed by the Sjögren's Tool for Assessing Response (STAR) | week 24
  STAR is a new response assessment tool for pSS including 5 aspects: systemic activity, patient-reported outcomes, lacrimal gland function, salivary gland function, and biomarkers, which can evaluate treatment response in all patients with pSS, including those with low systemic activity but high symptom burden.
  Response in system activity (3 points) is defined by a decrease of ≥3 in clinESSDAI and response in patient-reported outcome (3 points) is defined by a decrease of ≥1 point or 15% in ESSPRI. Response in lachrymal gland function (1 points) is assessed by Schirmer's test or ocular staining score. Response in Salivary gland function (1 points) was assessed by unstimulated whole salivary flow or ultrasound. Biological response (1 points) means decrease of serum IgG level ≥10% or decrease of RF level ≥25%. Candidate STAR responder is defined by total score of the above 5 domains ≥5.

SECONDARY OUTCOMES:
Change From Baseline in EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) Total Score during treatment | week 4, 12, 24, 52
  ESSDAI measures the disease activity of primary Sjögren's Syndrome from 12 aspects: constitutional, lymphadenopathy and lymphoma, glandular, articular, cutaneous, pulmonary, renal, muscular, peripheral nervous system, central nervous system, hematological, biological involvement. The score of each domain is obtained by multiplying the activity level by the domain weight, and the weight range is 1 to 6, and a numerical score is assigned according to the weight of each domain determined in advance. The sum of all single weighted domain scores is the total score, ranging from 0 ( best ) to 123 ( worst ). The higher the score, the stronger the disease activity. A clinically significant decrease ( ≥ 3 points ) compared with the baseline indicates an improvement in symptoms.
Change From Baseline in EULAR SS patient-reported index (ESSPRI) during treatment | week 4, 12, 24, 52
  ESSPRI was developed to assess patients' symptoms in primary Sjögren's Syndrome. It Includes three main symptoms, dryness, pain, and fatigue, and each with a score range of 0-10, and the ESSPRI score is the average of the three scores. A higher score indicated more severe symptoms.
Variation of lymphocyte subpopulations during the treatment of upadacitinib | week 4, 12, 24, 52
  Lymphocyte subgroups of T cell and B cell are analyzed during the treatment.
Alteration of inflammatory biomarkers and pathways after treatment of upadacitinib | week 4, 12, 24, 52
Change in quality of life(QOL) measured by 5-level EQ-5D version (EQ-5D-5L) compared with baseline | week 4, 12, 24, 52
  The EQ-5D-5L is a health-related quality-of-life instrument developed by the EuroQol Group. It is designed to measure health status across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Jing He, Principal Investigator — Peking University Institute of Rheuamotology and Immunology
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, China, China